CLINICAL TRIAL: NCT02137252
Title: Naltrexone Randomized Controlled Trial for Treatment-Emergent Fatigue in Patients Receiving Radiation Therapy for Breast Cancer
Brief Title: Naltrexone RCT for Treatment-Emergent Fatigue in Patients Receiving Radiation Therapy for Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: no enough patients
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Fremonta Meyer, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 14-056; R01CA150226 (NIH)
Record Dates: First submitted 2014-05-10; First posted 2014-05-13 (Estimated); Results first posted 2021-11-16 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Invasive Breast Cancer (Stage I-III); Ductal Carcinoma in Situ; Lobular Carcinoma in Situ; Lobular Carcinoma; Fatigue Related to Cancer Treatment
Keywords: Invasive Breast Cancer (Stage I-III); Ductal Carcinoma in Situ; Lobular Carcinoma in Situ; Lobular Carcinoma; Fatigue Related to Cancer Treatment
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ; Carcinoma, Lobular | interventions — Naltrexone; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naltrexone (Experimental): The treatment schedule includes a daily dose of naltrexone for 5 weeks. Treatment will be initiated at 25 mg/day during the first week to improve tolerability. The dose will be escalated to 50 mg/day after one week barring significant early improvement in fatigue or adverse events precluding dose escalation, and participants will continue to take 50 mg/day (or 25 mg/day if dose is not escalated) for 4 weeks to complete a 5-week treatment period.
  Interventions: Drug: Naltrexone
- Sugar Pill (Placebo Comparator): The treatment schedule includes a daily dose of equivalent placebo for 5 weeks. Treatment will be initiated at 25 mg/day during the first week to improve tolerability. The dose will be escalated to 50 mg/day after one week barring significant early improvement in fatigue or adverse events precluding dose escalation, and participants will continue to take 50 mg/day (or 25 mg/day if dose is not escalated) for 4 weeks to complete a 5-week treatment period.
  Interventions: Drug: Sugar Pill

INTERVENTIONS:
Drug: Naltrexone
  Other Names: ReVia®
  Arms: Naltrexone
Drug: Sugar Pill
  Arms: Sugar Pill

SUMMARY:
Naltrexone is a drug which blocks some effects of chemicals called beta-endorphins that are made in the body. Beta-endorphins can be made in response to stress, injury, and also pleasurable activities. In previous studies, it has been shown that levels of beta-endorphins in the blood go up during radiation therapy, and that this increase is linked to fatigue. This suggests that naltrexone may help to reduce fatigue in people who are getting radiation therapy In this research study, the investigators are looking to see whether naltrexone works better than a placebo in reducing fatigue during radiation therapy.

DETAILED DESCRIPTION:
This trial has two phases (a monitoring and an intervention phase).

Monitoring Phase: Prior to starting radiotherapy for non-metastatic breast cancer, participants will be approached and consented for the monitoring phase of the study, which involves longitudinal monitoring of fatigue in order to establish whether a patient develops fatigue after starting radiation. The level of pre-radiotherapy fatigue will be obtained during the final two weeks before radiotherapy is started. All participants will undergo weekly monitoring of fatigue via a brief self-report questionnaire. The monitoring period will continue up until one month after the conclusion of radiotherapy. Those whose fatigue symptoms increase above the pre-specified threshold at any point during the monitoring period will be approached about enrollment into the intervention phase of the study.

Intervention Phase: This is a randomized, double-blind, parallel-arm 5-week clinical trial which will be used to determine the effect of naltrexone on fatigue emerging during radiation therapy for non-metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria

Eligibility Criteria for Monitoring Phase

* Age ≥ 18
* Diagnosis of: invasive breast cancer (stage I-III), ductal carcinoma in situ, lobular carcinoma in situ, lobular carcinoma
* Plan to receive radiation therapy

Eligibility Criteria for Randomization Phase

* Participants may have had prior breast surgery and/or chemotherapy.
* Age ≥18 years.

  --Because no dosing or adverse event data are currently available on the use of naltrexone in cancer patients <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Participants must have acceptable pre-treatment laboratory values as defined below:

  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance ≥60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
  * If child-bearing potential, willingness to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document
* Receiving radiation therapy of any type at DFCI, BWH, or MGH (including but not limited to partial breast irradiation, two-field, three-field, and four-field plans)
* FACIT-F subscale score >=10 pre-radiation therapy and decrease in FACIT-F of 10 points or more as compared to pre-radiotherapy baseline

Exclusion Criteria:

Exclusion Criteria for Monitoring Phase

* Suicidal ideation, as determined via PHQ-9
* Non-English speaking

Exclusion Criteria for Randomization Phase

* Participants with major depressive disorder and/or suicidal ideation as determined by PHQ-9.
* Participants who are receiving any other investigational agents that might interact with study medication or influence the measurement of study outcomes.
* Participants with known metastatic disease should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to naltrexone.
* Participants who have used opioid-containing medications (including cough/cold medications containing codeine and/or antidiarrheals containing loperamide) in the past 2 weeks, or who are expected to require opioid-containing medications within the duration of the treatment period.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because naltrexone is category C agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with naltrexone, breastfeeding should be discontinued if the mother is treated with naltrexone.
* Participants using other contraindicated medications (thioridazine, yohimbine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-05; Primary Completion 2015-08-01 (Actual); Study Completion 2015-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fremonta Meyer, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hosptial, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the monitoring phase, eligibility for randomization was defined as FACIT-F subscale score >=10 pre-radiation therapy and decrease in FACIT-F of 10 points.
Groups:
- Naltrexone: The dose will be escalated to 50 mg/day (or equivalent placebo) after one week barring significant early improvement in fatigue or adverse events precluding dose escalation, and participants will continue to take 50 mg/day (or 25 mg/day if dose is not escalated) for 4 weeks to complete a 5-week treatment period.
- Sugar Pill: daily dose placebo for 5 week treatment period
Period: Overall Study
Arm/Group | Naltrexone | Sugar Pill
Started (Represents intervention phase) | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — trial terminated early | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Sugar Pill: daily dose placebo for 5 week treatment period
- Total: Total of all reporting groups
Arm/Group | Naltrexone | Placebo: Sugar Pill | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Mean (Full Range); unit: Years] | 49 [42 to 56] | 59 [59 to 59] | 52.3 [41 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in FACIT-fatigue Subscale Score From Randomization to End of Study
Description: Functional Assessment of Chronic Illness Therapy-Fatigue Subscale (FACIT-fatigue subscale): This 13-item self-report scale measuring fatigue and functional impairment as a result of fatigue has been validated in cancer patients (Cella et al. Cancer 2002;94:528-38) The scale is reverse-scored and the range is 0 (maximum fatigue) - 52 (minimum fatigue). According to ICD10 criteria, a score <= 34 indicates significant cancer related fatigue. A change of 10 points has been shown to constitute a clinically meaningful difference on this subscale.
Time Frame: Evaluated at baseline, weekly monitoring visits from start of radiation therapy and meets fatigue eligibility threshold
Population: trial terminated early
Groups:
- Naltrexone: The treatment schedule includes a daily dose of naltrexone for 5 weeks. Treatment will be initiated at 25 mg/day during the first week to improve tolerability. The dose will be escalated to 50 mg/day after one week barring significant early improvement in fatigue or adverse events precluding dose escalation, and participants will continue to take 50 mg/day (or 25 mg/day if dose is not escalated) for 4 weeks to complete a 5-week treatment period.
  Naltrexone
- Sugar Pill: The treatment schedule includes a daily dose of equivalent placebo for 5 weeks. Treatment will be initiated at 25 mg/day during the first week to improve tolerability. The dose will be escalated to 50 mg/day after one week barring significant early improvement in fatigue or adverse events precluding dose escalation, and participants will continue to take 50 mg/day (or 25 mg/day if dose is not escalated) for 4 weeks to complete a 5-week treatment period.
  Sugar Pill
Arm/Group | Naltrexone | Sugar Pill
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants in the monitoring phase of the study will be followed for a maximum of 10 weeks, ending 4 weeks after cessation of radiotherapy or until they consent (if eligible) to participate in the intervention phase of the study, followed until the end of the study and beyond, until resolution or stabilization of the adverse event has occurred.
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Arm/Group | Naltrexone | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Naltrexone (N=2) | Sugar Pill (N=1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 | 1
fatigue (General disorders) | 2 | 1
headache (Nervous system disorders) | 1 | 0
nausea (Gastrointestinal disorders) | 1 | 0
dizziness (Gastrointestinal disorders) | 1 | 1
irritability (General disorders) | 1 | 1
mental fogginess (Nervous system disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-03-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT02137252/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan (2016-03-30): https://cdn.clinicaltrials.gov/large-docs/52/NCT02137252/Prot_SAP_001.pdf